CLINICAL TRIAL: NCT05979363
Title: Safety and Efficiency of VRd Combining BCMA CAR-T Regimen for Transplant-ineligible Patients With Primary Plasma Cell Leukemia: a Prospective, Single-arm, Single-center, Phase II Study.
Brief Title: A Study of Bortezomib, Lenalidomide and Dexamethasone (VRd)-Based Regimen Followed by BCMA CAR-T Therapy in Transplant-Ineligible Patients With Primary Plasma Cell Leukemia
Acronym: CAREMM-002
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023034
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Plasma Cell Leukemia
MeSH Terms: conditions — Leukemia, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VRD-based Regimen Combined With BCMA CART (Experimental): VRD：Bortezomib, Lenalidomide and Dexamethasone Bortezomib SC 1.3mg/sqm on day 1,8,15,22, Lenalidomide oral 25 mg on day 1-21, and Dexamethasone 40mg on day 1,8,15,22 in a 28-day cycle.
  Autologous BCMA-directed CAR-T cells, infusion intravenously at a target dose of 2-4 x 10^6 anti-BCMA CAR+T cells/kg.
  Participants will receive VRD-based induction, BCMA CAR-T infusion, VR consolidation, VR maintenance.
  Interventions: Biological: anti-BCMA CAR-T; Drug: VRD-based regimen

INTERVENTIONS:
Biological: anti-BCMA CAR-T — Autologous BCMA-directed CAR-T cells, infusion intravenously at a target dose of 2.0-4.0 x 10^6 anti-BCMA CAR+T cells/kg.
Drug: VRD-based regimen — Bortezomib, Lenalidomide and Dexamethasone

SUMMARY:
This is a single-arm, open-label study to evaluate the efficacy and safety of VRD-based regimen combined with BCMA CAR-T in transplant-ineligible patients with primary plasma cell leukemia

DETAILED DESCRIPTION:
The study is a prospective, single-arm, single-centre, phase II study designed to evaluate the efficacy and safety of treatment with VRD-based regimen combined with BCMA CAR-T in transplant-ineligible patients with primary plasma cell leukemia. Patients received 3 courses of induction therapy with VRD-based regimen followed by infusion of BCMA CAR-T cells. Patients then received 3 courses of VR consolidation therapy, followed by VR maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years.
2. Participants with documented primary plasma cell leukemia according to IMWG diagnostic criteria (circulating plasma cells ≥5%, determined by morphology on peripheral blood smear; or absolute value of peripheral blood tumorigenic plasma cells exceeds 2×10^9/L).
3. Measurable disease, at screening as defined by any of the following: Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or Light chain MM without measurable disease in serum or urine: serum Ig free-light chain (FLC) ≥10 mg/dL and abnormal serum Ig kappa lambda FLC ratio.
4. Not considered for high-dose chemotherapy with Autologous Stem Cell Transplant (ASCT) due to: Ineligible due to advanced age (≥65); or Ineligible evaluated by researchers; or Eastern Cooperative Oncology Group Performance Status grade of 3 or 4; or Repeated hematopoietic stem cell mobilization failure； or Deferral of high-dose chemotherapy with ASCT as initial treatment.
5. Bone marrow sample is confirmed as BCMA-positive by flow cytometry or pathological examination.
6. All screening blood biochemistry: tests should be performed according to the protocol and within 14 days before enrollment. Screening laboratory values must meet the following criteria: a.TBIL<2 x upper limit of normal (ULN) (<3 x ULN in patients with Gilbert's syndrome); b.AST and ALT <3 x ULN.; c. Creatinine clearance ≥ 30mL/min (calculated using Cockroft-Gault formula).
7. Routine blood tests (performed within 7 days, no RBC transfusion, no G-CSF/GM-CSF/platelet agonists, no drug correction within 14 days before screening, no PLT transfusion within 7 days) : WBC ≥ 1.5 x 109/L, ANC ≥ 1.0 x 109/L, Hb ≥ 70 g/L PLT ≥ 75 x 109/L (if BMPC < 50%) or PLT ≥ 50 x 109/L (if BMPC ≥ 50%).
8. Patients must be able to take prophylactic anticoagulant therapy as recommended by the study.
9. The woman is not breastfeeding, is not pregnant and agrees not to be pregnant during the study period and for the following 12 months. Male patients agreed that their spouse would not become pregnant during the study period and for 12 months thereafter.

Exclusion Criteria:

1. Documented active amyloidosis.
2. Documented with central nervous system (CNS) invasion.
3. Prior exposure to any BCMA-targeted therapy or CAR-T therapy.
4. Patients with peripheral neuropathy greater than grade 2 or peripheral neuropathy greater than grade 2 with pain at baseline, regardless of whether they were currently receiving medical therapy.
5. Known intolerance, hypersensitivity, or contraindication to glucocorticoids, bortezomib, lenalidomide, and BCMA-CART cellular products.
6. Seropositive for human immunodeficiency virus (HIV)
7. Hepatitis B infection
8. Hepatitis C infection
9. Life expectancy of <6 months
10. Women who are pregnant or breastfeeding
11. Any active gastrointestinal dysfunction that affects the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that may affect the absorption of the studied treatment medication
12. Subjects had major surgery within 2 weeks before randomization (for example, general anesthesia), or is not fully recovered from the surgery, or surgery is arranged during study period.
13. Received live attenuated vaccine within 4 weeks prior to study treatment.
14. According to the researcher's judgment, any condition including but not limited to serious mental illness, medical illness, or other symptoms/conditions that may affect study treatment, compliance, or the capability of providing informed consent.
15. Necessary medication or supportive therapy is contraindicated with study treatment.
16. Any diseases or complications that may interfere with the study.
17. Patients are not willing to or cannot comply with study scheme.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 2 year
  The incidence of treatment-emergent adverse events (TEAEs)
MRD-negative rate | within 1 week after consolidation treatment
  achieving MRD-negative, as determined by NGS/NGF after consolidation treatment

SECONDARY OUTCOMES:
Complete response rate (CRR) | within 1 week after induction therapy, 1 month after the CAR-T cell transfusion, within 1 week after consolidation therapy
  CR or better is defined as percentage of participants who achieve a CR response or Stringent Complete Response (sCR) response accoording to the IMWG criteria
Progression free survival (PFS) | Up to 2 year
  Progression free survival is defined as the time from the date of diagnosis to the date of first documented PD, as defined in the IMWG criteria, or death due to any cause, whichever occurs first
Overall Survival (OS) | Up to 5 year
  Overall survival is measured from the date of diagnosis to the date of the participant's death.
Duration of Remission(DOR) | Up to 2 year
  Duration from the first evaluation of at least partial remission (PR) to the onset of disease progression or death due to disease progression (whichever occurs first)

OTHER OUTCOMES:
The duration of CART cell in vivo | Up to 1 year
  The copies of BCMA-CART DNA in peripheral blood with qPCR method
Change from Baseline in Physical status assessed by International Myeloma Working Group Comprehensive Geriatric Assessment (IMWG-CGA) scores | Baseline up to 5 years
  The IMWG-CGA was calculated by combining age, activities of daily living (ADL), instrumental ADL (IADL), and Charlson Comorbidity Index (CCI), which ranges from 0 to 5 with higher scores indicating worse physical condition and greater weakness.
Change from Baseline in Physical status assessed by activities of daily living (ADL) scores | Baseline up to 5 years
  The ADL includes 4 items (transfer, bed mobility, toileting, and eating), which range from 0 to 6 scores. A higher score represents worse physical condition and greater weakness.
Change from Baseline in Physical status assessed by instrumental activities of daily living (IADL) scores | Baseline up to 5 years
  The IADL includes 5 items (cooking, cleaning, transportation, laundry, and managing finances), which range from 0 to 8 scores. A higher score represents worse physical condition and greater weakness.
Change from Baseline in Physical status assessed by Charlson Comorbidity Index (CCI) | Baseline up to 5 years
  The CCI estimates the number and the severity of comorbidities, including nineteen diseases with a score varying from 1 to 6 for each of them in accordance to their severity. The score can range from 0 to 37. A higher score represents more severe comorbidities.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No